CLINICAL TRIAL: NCT01216397
Title: Relative Bioavailability of Two Different Batches of a 2.5 mg Linagliptin / 1000 mg Metformin Fixed Dose Combination Tablet (FDC) in Healthy Male and Female Volunteers (an Open-label, Randomised, Single Dose, Two-way Crossover, Phase I Trial)
Brief Title: Relative Bioavailability of Two Different Batches of a Linagliptin / Metformin Combination Tablet in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1288.6; 2010-019291-75 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-10-04; First posted 2010-10-07 (Estimated); Results first posted 2012-04-25 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin; Metformin

ARMS (2):
- Linagliptin/Metformin (standard batch) (Experimental): Fixed dose combination tablet
  Interventions: Drug: Linagliptin/Metformin (standard batch)
- Linagliptin/Metformin (side batch) (Experimental): Fixed dose combination tablet
  Interventions: Drug: Linagliptin/Metformin (side batch)

INTERVENTIONS:
Drug: Linagliptin/Metformin (standard batch) — Fixed dose combination tablet
  Arms: Linagliptin/Metformin (standard batch)
Drug: Linagliptin/Metformin (side batch) — Fixed dose combination tablet
  Arms: Linagliptin/Metformin (side batch)

SUMMARY:
The objective of the current study is to investigate the relative bioavailability of two different batches of a 2.5 mg linagliptin / 1000 mg metformin fixed dose combination tablet (FDC).

ELIGIBILITY:
Inclusion criteria:

1. Healthy males and females according to the following criteria: Based upon a complete medical history, including physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), clinical laboratory tests
2. Age 21 to 50 years (incl.)
3. Body Mass Index (BMI) 18.5 to 29.9 kg/m2 (incl.)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion criteria:

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells or blackouts
7. Chronic or relevant acute infections
8. History of relevant allergy or hypersensitivity (including allergy to drug or its excipients)
9. Intake of drugs within one month or less than 10 half-lives of the respective drug prior to first study drug administration
10. Participation in another trial with an investigational drug within 2 months prior to administration or during the trial
11. Smoker (more than 10 cigarettes or 3 cigars 3 pipes daily)
12. Alcohol abuse (average consumption of more than 20 g/day in females and 30 g/day in males)
13. Drug abuse
14. Blood donation (more than 100 mL within four weeks prior to day 1 of visit 2)
15. Any laboratory value outside the reference range that is of clinical relevance
16. Inability to comply with dietary regimen of trial site

    For female subjects of childbearing potential only:
17. Positive pregnancy test, pregnancy or planning to become pregnant 1 month before study or within 2 months after study completion
18. No adequate contraception 1 month before study and until 2 month after study completion, e.g. not any of the following: implants, injectables, combined hormonal contraceptives, hormonal IUD (intrauterine device), sexual abstinence for at least 1 month prior to first study drug administration, vasectomised partner (vasectomy performed at least 1 year prior to enrolment), or surgical sterilisation (including hysterectomy). Females, who do not have a vasectomised partner, are not sexually abstinent or surgically sterile will be asked to use an additional barrier method (e.g. condom).
19. Lactation

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1288.6.1 Boehringer Ingelheim Investigational Site, Ingelheim, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an open-label, single-dose, randomised, 2-way crossover trial. Subjects were equally randomised to one of two sequences, and in general terms, AB or BA. Hence, 20 subjects were in group AB and 20 in group BA. All 40 subjects received A and B. The numbers presented in the milestones are overall, which is consistent with the trial report.
Groups:
- Standard Batch Then Side Batch: Linagliptin/metformin FDC tablet from standard batch, then Linagliptin/metformin FDC tablet from side batch
- Side Batch Then Standard Batch: Linagliptin/metformin FDC tablet from side batch, then Linagliptin/metformin FDC tablet from standard batch
Period: Period 1
Arm/Group | Standard Batch Then Side Batch | Side Batch Then Standard Batch
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Washout (35 Days)
Arm/Group | Standard Batch Then Side Batch | Side Batch Then Standard Batch
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Standard Batch Then Side Batch | Side Batch Then Standard Batch
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Treatment with standard batch and side batch
Arm/Group | All Participants
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.8 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 20
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 23.74 (2.74)

OUTCOME MEASURES:

1. Primary Outcome: Linagliptin: Maximum Measured Concentration (Cmax)
Description: Geometric mean of Cmax of Linagliptin
Time Frame: Day 1 to 35 for period 1, and Day 36 to 70 for period 2
Population: Treated Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- Standard Batch: standard batch of a 2.5 mg linagliptin/ 1000mg metformin FDC
- Side Batch: side batch of a 2.5 mg linagliptin/ 1000mg metformin FDC
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
nmol/L | 5.36 (20.3) | 5.39 (20.3)
Statistical Analysis 1: Comparison: Standard Batch vs Side Batch; Standard batch vs. Side batch; Test type: Superiority or Other; ANOVA; adjusted gMean ratio = 99.4, 90% CI [94.2 to 105.0]

2. Primary Outcome: Area Under the Concentration-time Curve of Linagliptin in Plasma Over the Time Interval 0 to 72 Hours (AUC0-72)
Description: Geometric mean of AUC0-72 of Linagliptin
Time Frame: Day 1 to 35 for period 1, and Day 36 to 70 for period 2
Population: Treated Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*hr/L
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
nmol*hr/L | 179 (21.6) | 179 (20.5)
Statistical Analysis 1: Comparison: Standard Batch vs Side Batch; Standard batch vs. Side batch; Test type: Superiority or Other; ANOVA; adjusted gMean ratio = 100.1, 90% CI [96.1 to 104.2]

3. Secondary Outcome: Linagliptin: AUC0-infinity
Description: Geometric mean of AUC0-infinity of Linagliptin
Time Frame: Day 1 to 35 for period 1, and Day 36 to 70 for period 2
Population: Treated Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*hr/L
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
nmol*hr/L | 267 (25.4) | 267 (23.6)
Statistical Analysis 1: Comparison: Standard Batch vs Side Batch; Standard batch vs. Side batch; Test type: Superiority or Other; ANOVA; adjusted gMean ratio = 100.1, 90% CI [94.7 to 105.8]

4. Secondary Outcome: Linagliptin: Percentage of AUCtz-∞ Obtained by Extrapolation
Description: Geometric Mean of percentage of AUCtz-∞ of linagliptin, where percentage is the unit of measurement.
Time Frame: Day 1 to 35 for period 1, and Day 36 to 70 for period 2
Population: Treated Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
percentage | 32.6 (17.5) | 32.1 (20.3)

5. Secondary Outcome: Linagliptin: Time to Maximum Measured Concentration of the Analyte in Plasma (Tmax)
Description: Median of the t_max of linagliptin
Time Frame: Day 1 to 35 for period 1, and Day 36 to 70 for period 2
Population: Treated Set
Measure: Median (Full Range); unit: hr
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
hr | 3.00 [0.667 to 6.02] | 3.00 [0.983 to 6.02]

6. Secondary Outcome: Linagliptin: λz (Terminal Elimination Rate Constant in Plasma)
Description: Geometric mean of the λ_z of linagliptin
Time Frame: Day 1 to 35 for period 1, and Day 36 to 70 for period 2
Population: Treated Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hr
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
1/hr | 0.0153 (17.1) | 0.0152 (21.6)

7. Secondary Outcome: t1/2 (Terminal Half-life of the Analyte in Plasma)
Description: Geometric mean of the t1/2 of linagliptin
Time Frame: Day 1 to 35 for period 1, and Day 36 to 70 for period 2
Population: Treated Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
hr | 45.4 (17.1) | 45.6 (21.6)

8. Secondary Outcome: Linagliptin: MRTpo (Mean Residence Time of the Analyte in the Body After Peroral Administration)
Description: Geometric mean of the MRTpo of linagliptin
Time Frame: Day 1 to 35 for period 1, and Day 36 to 70 for period 2
Population: Treated Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
hr | 64.6 (15.7) | 64.5 (19.5)

9. Secondary Outcome: Linagliptin: Apparent Clearance of the Analyte in Plasma After Extravascular Administration (CL/F)
Description: Geometric mean of the CL/F of linagliptin
Time Frame: Day 1 to 35 for period 1, and Day 36 to 70 for period 2
Population: Treated Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
mL/min | 330 (25.4) | 330 (23.6)

10. Secondary Outcome: Linagliptin: Apparent Volume of Distribution During the Terminal Phase Following an Extravascular Dose (Vz/F)
Description: Geometric mean of the Vz/F of linagliptin
Time Frame: Day 1 to 35 for period 1, and Day 36 to 70 for period 2
Population: Treated Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
Liter | 1300 (22.8) | 1300 (24.6)

11. Primary Outcome: Metformin: Cmax
Description: Geometric Mean of Cmax of Metformin
Time Frame: Day 1 to 35 for period 1, and Day 36 to 70 for period 2
Population: Treated Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
ng/mL | 1790 (23.0) | 1820 (25.5)
Statistical Analysis 1: Comparison: Standard Batch vs Side Batch; Standard batch vs. Side batch; Test type: Superiority or Other; ANOVA; adjusted gMean ratio = 97.9, 90% CI [92.5 to 103.7]

12. Primary Outcome: Metformin: AUC0-tz
Description: Geometric Mean of AUC0-tz of Metformin
Time Frame: Day 1 to 35 for period 1, and Day 36 to 70 for period 2
Population: Treated Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
ng*hr/mL | 12100 (21.4) | 12100 (19.4)
Statistical Analysis 1: Comparison: Standard Batch vs Side Batch; Test type: Superiority or Other; ANOVA; adjusted gMean ratio = 100.4, 90% CI [95.7 to 105.4]

13. Secondary Outcome: Metformin: AUC0-infinity
Description: Geometric Mean of AUC0-infinity of Metformin
Time Frame: Day 1 to 35 for period 1, and Day 36 to 70 for period 2
Population: Treated Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
ng*h/mL | 12400 (21.2) | 12300 (19.9)
Statistical Analysis 1: Comparison: Standard Batch vs Side Batch; Standard batch vs. Side batch; Test type: Superiority or Other; ANOVA; adjusted gMean ratio = 100.3, 90% CI [95.7 to 105.2]

14. Secondary Outcome: Metformin: Percentage of AUCtz-∞ Obtained by Extrapolation
Description: Geometric Mean of the percentage of AUCtz-infinity of Metformin, where percentage is the unit of measurement.
Time Frame: Day 1 to 35 for period 1, and Day 36 to 70 for period 2
Population: Treated Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
percentage | 1.51 (87.4) | 1.52 (97.0)

15. Secondary Outcome: Metformin: Tmax
Description: Median of tmax of metformin
Time Frame: Day 1 to 35 for period 1, and Day 36 to 70 for period 2
Population: Treated Set
Measure: Median (Full Range); unit: hr
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
hr | 1.99 [0.667 to 4.02] | 2.00 [0.65 to 4.02]

16. Secondary Outcome: Metformin: λz (Terminal Elimination Rate Constant in Plasma)
Description: Geometric mean of λz of metformin
Time Frame: Day 1 to 35 for period 1, and Day 36 to 70 for period 2
Population: Treated Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hr
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
1/hr | 0.0493 (71.0) | 0.0514 (84.3)

17. Secondary Outcome: Metformin: t1/2 (Terminal Half-life of the Analyte in Plasma)
Description: Geometric mean of t1/2 of metformin
Time Frame: Day 1 to 35 for period 1, and Day 36 to 70 for period 2
Population: Treated Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
hr | 14.1 (71.0) | 13.5 (84.3)

18. Secondary Outcome: Metformin: MRTpo (Mean Residence Time of the Analyte in the Body After Peroral Administration)
Description: Geometric mean of MRTpo of metformin
Time Frame: Day 1 to 35 for period 1, and Day 36 to 70 for period 2
Population: Treated Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
hr | 8.27 (31.1) | 8.23 (36.9)

19. Secondary Outcome: Metformin: CL/F
Description: Geometric mean of CL/F of metformin
Time Frame: Day 1 to 35 for period 1, and Day 36 to 70 for period 2
Population: Treated Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
mL/min | 1350 (21.2) | 1350 (19.9)

20. Secondary Outcome: Metformin: Vz/F
Description: Geometric mean of Vz/F of metformin
Time Frame: Day 1 to 35 for period 1, and Day 36 to 70 for period 2
Population: Treated Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
Liter | 1640 (74.3) | 1580 (82.4)

21. Secondary Outcome: Electrocardiogram (ECG), Vital Signs, Physical Finding or Laboratory Finding Abnormalities
Description: 12-lead-Electrocardiogram (ECG), vital sign (blood pressure and pulse rate), physical finding and laboratory abnormalities
Time Frame: Day 1 to 4 for period 1, and day 36 to 39 for period 2
Population: Treated Set
Measure: Number; unit: Participants
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
Participants
  Physical examination abnormalities | 0 | 0
  Vital sign abnormalities | 0 | 0
  ECG abnormalities | 0 | 0
  Laboratory finding abnormalities | 0 | 0

22. Secondary Outcome: Participants With Treatment Emergent Adverse Events
Description: Number of patients with treatment emergent AEs
Time Frame: Day 1 to 4 for period 1, and day 36 to 39 for period 2
Population: Treated Set
Measure: Number; unit: Participants
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
Participants
  Headache | 6 | 9
  Nausea | 0 | 1
  Vomiting | 2 | 1
  Fatigue | 1 | 0

23. Secondary Outcome: Participants Who Discontinued the Trial Because of an Adverse Event
Description: Number of participants who discontinued the trial because of an adverse event
Time Frame: Day 1 to 4 for period 1, and day 36 to 39 for period 2
Population: Treated Set
Measure: Number; unit: Participants
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
Participants | 0 | 0

24. Secondary Outcome: Assessment of Tolerability by the Investigator
Description: Qualitative variable assessing the tolerability by the investigator
Time Frame: Day 1 to 4 for period 1, and day 36 to 39 for period 2
Population: Treated Set
Measure: Number; unit: Participants
Arm/Group | Standard Batch | Side Batch
Number analyzed (Participants) | 40 | 40
Participants
  Good | 39 | 40
  Not satisfactory | 1 | 0

ADVERSE EVENTS:
Time Frame: 4 days (period 1) + 4 days (treatment period 2)
Description: Two identical treatment periods with an interval of at least 35 days between drug administrations.
Arm/Group | Standard Batch | Side Batch
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 7/40 | 11/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Batch (N=40) | Side Batch (N=40)
Headache (Nervous system disorders) | 7 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.